CLINICAL TRIAL: NCT00935831
Title: A Phase I, Single-Dose, Randomized and Single-Blind (Part 1), Fixed Sequence and Open-Label (Part 2), Studyto Evaluate the Safety, Pharmacokinetics, andPharmacodynamics of 1278863A in Subjects With RenalImpairment and Matched Healthy Volunteers
Brief Title: Single Dose Safety Study for Compound to Treat Anemia in Patients With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 112843
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Kidney Disease
Keywords: Tolerability; Safety; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Subjects with renal impairment, non-dialysis (Experimental): Subjects with moderate to severe renal impairment equivalent to National Kidney Foundation Kidney Disease Outcomes Quality Initiative stage 3 and stage 4 who are not undergoing dialysis will be included. Subjects will receive single 50 mg and 150 mg oral doses of GSK1278863A across two dosing periods in a single-blind, randomized sequence. Doses of GSK1278863A will be given as 25 mg and 100 mg tablets, with matching placebo tablets to maintain treatment blinding.
  Interventions: Drug: GSK1278863A; Drug: Placebo
- Healthy volunteers (Experimental): Healthy subjects will be matched to the moderate and severe renally impaired subjects for gender, age, and BMI. Subjects will receive single 50 mg and 150 mg oral doses of GSK1278863A across two dosing periods in a single-blind, randomized sequence. Doses of GSK1278863A will be given as 25 mg and 100 mg tablets, with matching placebo tablets to maintain treatment blinding.
  Interventions: Drug: GSK1278863A; Drug: Placebo
- Hemodialysis dependent subjects (Experimental): The arm will consist of subjects with severe renal impairment (end-stage renal failure) who have been on stable hemodialysis treatment scheduled three times per week. Subjects will receive single oral doses of 150 mg GSK1278863A in each of 2 dosing periods in an open-label, fixed sequence. GSK1278863A will be administered just prior to receiving scheduled hemodialysis in Dosing Period 1. In Dosing Period 2, subjects will receive a single oral dose of GSK1278863 the morning after completion of a scheduled hemodialysis session.
  Interventions: Drug: GSK1278863A

INTERVENTIONS:
Drug: GSK1278863A — 50mg, 150mg
Drug: Placebo — matching placebo
  Arms: Healthy volunteers; Subjects with renal impairment, non-dialysis

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of single doses of compound 1278863A in subjects with renal impairment.

DETAILED DESCRIPTION:
Compound 1278863A is a novel small molecule agent, which stimulates erythropoiesis through inhibition of hypoxia-inducible factor (HIF)-prolyl hydroxylases (EGLNs). This compound is being developed for the treatment of anemia. This study, PHI112843, will be the first administration of 1278863A to investigate the safety, tolerability, pharmacokinetics and/or pharmacodynamics of single oral doses of 50 mg and 150 mg in pre-dialysis subjects with moderate or severe renal impairment and 150 mg in hemodialysis-dependent subjects. Four to eight subjects will complete each dose cohort. Multiple blood samples for pharmacokinetic and/or pharmacodynamic analyses will be obtained post-dose in each cohort. Safety will be assessed by measurement of vital signs, cardiac monitoring, collection of adverse event assessments and laboratory safety tests.

ELIGIBILITY:
Inclusion Criteria:

1. A male or female is eligible to enroll and participate in this study if he/she:

   * (Part 1) has Moderate to Severe Renal Impairment (equivalent to NKF KDOQI Stage 3 or 4, not receiving dialysis) as determined by estimated Glomerular Filtration Rate (eGFR) calculated by the abbreviated MDRD equation, OR has Normal Renal Function determined by creatinine clearance (CLCR) via the Cockcroft-Gault equation, using serum creatinine and demographic data, obtained at Screening. Subjects with Normal Renal Function should have no greater than trace blood or protein on Screening urinalysis.
   * (Part 2) has severe renal impairment (end-stage renal failure) and has been on stable hemodialysis treatment (three times weekly) for 3 months prior to Screening.
   * otherwise healthy or considered clinically stable with respect to underlying renal impairment as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
   * has clinical laboratory test results that are considered clinically stable in the opinion of the Principal Investigator, especially if the clinical abnormality or laboratory parameter is deemed associated with the subject's underlying renal impairment. A normal subject with a clinical abnormality or laboratory parameters outside the reference range may be included only if the Investigator and the Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
2. Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
3. A female subject is eligible to participate if she is of:

   - Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods described in the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT.

   Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
4. Male subjects must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study drug until completion of the Follow-up visit.
5. Body weight greater than or equal to 50 kg and BMI within the range 17 - 33 kg/m2 (inclusive).
6. AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
7. QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block. These can be based on single ECG value or average of triplicate values obtained over brief recording period.
8. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. A hemoglobin value at Screening is:

   * Healthy male subjects or post-menopausal females: > 16.5 g/dL
   * Healthy female subjects: > 15.5 g/dL
   * Renally impaired male or female subjects: <10 g/dL
2. The values of hematological parameters at Screening, for healthy subjects only, are outside the reference range and clinically significant deemed by the Investigator and Medical Monitor
3. The values of the following tests at Screening, for healthy subjects only, are:

   * TIBC: outside the reference range
   * Serum iron: outside the reference range
   * Serum ferritin: outside the reference range
4. Clinically significant abnormal CPK determined by the Investigator and Medical Monitor.
5. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of Screening.
6. A positive test for HIV antibody.
7. A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines. A positive pre-study drug screen, for medications that are prescribed to a subject for pre-existing condition(s), may be allowed if in the opinion of the Investigator and Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
8. History of drug abuse or dependence within 6 months of the study.
9. History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
10. History of regular use of tobacco- or nicotine-containing in excess of 10 cigarettes per day or equivalent and an inability to abstain from tobacco or nicotine use from admission to the clinical research unit until discharge for each dosing period.
11. Use of prescription medication known to be inhibitors of BCRP.
12. Use of non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study drug, unless in the opinion of the Investigator and Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
13. History of sensitivity to any of the study drugs, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
14. History of sensitivity to heparin or heparin-induced thrombocytopenia. (if the clinical research unit uses heparin to maintain intravenous cannula patency)
15. Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, and/or hepatic function that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Examples of conditions that could interfere with normal gastrointestinal anatomy or motility include cholecystectomy, gastrointestinal bypass surgery, partial or total gastrectomy, small bowel resection, vagotomy, malabsorption, Crohn's disease, ulcerative colitis, or celiac sprue. Examples of conditions that could interfere with hepatic function include Gilberts syndrome.
16. History of peptic ulcer disease.
17. Subjects with polycystic kidney disease.
18. Post-renal transplantation subjects.
19. History of malignancy tumor. Non-melanoma skin cancer that has been definitely removed is allowed.
20. Pregnant females as determined by positive serum Beta-hCG test at Screening or prior to dosing.
21. Lactating females.
22. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
23. Unwillingness or inability to follow the procedures, or lifestyle and/or dietary restrictions outlined in the protocol.
24. Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices of the prohibited fruits from 7 days prior to the first dose of study drug in Dosing Period 1 until the collection of the final pharmacokinetic blood sample in Dosing Period 2, unless in the opinion of the Investigator and Medical Monitor this will not interfere with the study procedures or compromise subject safety.
25. The subject has participated in a clinical trial and has received an experimental investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
26. Exposure to more than four experimental investigational products within 12 months prior to the first dosing day.
27. Subject is mentally or legally incapacitated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-08-12 (Actual); Primary Completion 2010-04-27 (Actual); Study Completion 2010-04-27 (Actual)

PRIMARY OUTCOMES:
AUC (0-24), Cmax, tmax and half-life | Parts 1&2: Days 1-3

SECONDARY OUTCOMES:
Adverse Events reporting | throughout study
Safety Labs (Chemistry) | Screening, Day -1, 2, 3
Safety Labs (Hematology) | Screening, Days -1, 2, 3
Safety Labs (Urinalysis) | Screening, Days -1, 2, 3
Vital Signs (blood pressure and heart rate) | Screening, Days 1, 2, 3
12-lead ECG | Screening, Day 1
Clinical Monitoring/Observation | throughout
Actual values, rate of rise, rate of decline and maximum change from baseline in erythropoietin | Days 1, 2, 3
Actual values, rate of rise, rate of decline and maximum change from baseline in VEGF | Days 1, 2
Actual values, rate of rise, rate of decline and maximum change from baseline in Hepcidin | Days 1, 2
Actual values, rate of rise, rate of decline and maximum change from baseline in TIBC (total iron binding capacity) | Screening, Days 1, 3

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Christchurch, New Zealand

REFERENCES:
- See also: Results for study 112843 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112843?search=study&search_terms=112843#rs